CLINICAL TRIAL: NCT06556095
Title: Histologic Evaluation of Wound Healing After Ridge Preservation Using Allograft Hydrated With Dexamethasone Versus Saline
Brief Title: Ridge Preservation With FDBA (Freeze Dried Bone Allograft) Using Dexamethasone vs. Saline
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000655
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bone Graft; Tooth Extraction
Keywords: Allograft; Ridge preservation; Dexamethasone
MeSH Terms: interventions — Dexamethasone; Solutions

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial examining wound healing after tooth extraction and ridge preservation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be 1:1 so that 22 subjects are enrolled in each group (test and control). Patients will be blind to the hydrating solution used for their bone graft. Histomorphometric examiners will be blinded when the bone cores are evaluated for % vital bone, % residual graft and % CT/other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ridge preservation test group (Experimental): Patients will be randomized to one of the experimental treatment group immediately following tooth extraction and debridement of the socket (test: hydration of allograft with 4mg/1ml dexamethasone solution)
  Interventions: Drug: Dexamethasone 4mg/ml solution
- Ridge preservation control group (No Intervention): Patients will be randomized to the control group immediately following tooth extraction and debridement of the socket (control: hydration of allograft with normal saline solution)

INTERVENTIONS:
Drug: Dexamethasone 4mg/ml solution — The study intervention dexamethasone solution (4mg/ml) is used to hydrate bone allograft.
  Other Names: Dexamethasone
  Arms: Ridge preservation test group

SUMMARY:
Following the removal of a tooth, a bone graft is often placed in the socket to try to maintain the volume of bone that was there when the tooth was present so that the bone does not "shrink". The bone graft is kept in place with a small piece of material over the top of the tooth socket and with stitches. This procedure is called "Ridge Preservation". Many different materials are used for ridge preservation, including bone allografts (bone grafts derived from a human tissue donor). These bone allografts are dehydrated (dried) during processing. Before using the material in the socket, the material is re-hydrated (wetted). The most common hydrating (wetting) agent is normal saline (sterile salt water), but other hydrating agents such as blood can also be used. The bone allograft used in this study is Food and Drug Administration (FDA) approved.

DETAILED DESCRIPTION:
In this study, the investigators are examining if there is any difference in new bone formation in the tooth socket when the bone allograft placed after tooth extraction is hydrated with a solution of dexamethasone rather than normal saline. Dexamethasone is a steroid that is used routinely in medicine and dentistry as an inflammatory medication which can decrease things like swelling or pain. In this study, after removing the tooth the bone allograft will be hydrated in either saline or dexamethasone solution and then placed into the socket. After healing, a dental implant will later be placed at the same site. The graft material is used as part of standard care in dental practices, but it is not clear if the healing following use of allograft hydrated in dexamethasone is similar or different to hydrating with saline.

At the end of this study the researchers hope to learn the following: How much new bone formation occurs inside the tooth socket at approximately 16 weeks of healing after ridge preservation with allograft hydrated in either saline or dexamethasone solution?

This will be done by examining the bone retrieved from the implant site during the placement of the implant at study visit #5. This bone is normally removed during the drilling of the implant site and discarded as part of standard care. As part of this study, the bone specimen will be removed as normal but will not be discarded; instead, it will be analyzed for the purpose of this research study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 to 89
* One tooth, excluding molars, that has been identified by dental faculty as requiring a single tooth extraction
* A dental implant is indicated and treatment planned to replace the missing tooth
* Site has adequate restorative space for a dental implant-retained restoration
* Site has at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Site has a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
* Patients are nonsmokers or former smokers. Current smokers may be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Patient allergic to dexamethasone
* Will not cooperate with the follow-up schedule.
* Patients will not be entered who are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period (as confirmed verbally; an over-the-counter pregnancy test will be provided if pregnancy status is unknown or suspected). Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
* Smokers who smoke >10 cigarettes per day
* Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Bone Formation | Baseline to 16 weeks (±2 weeks)
  Difference in percentage of new bone formation at 16 weeks (±2 weeks) after ridge preservation is performed using a combination freeze-dried bone allograft (70% mineralized FDBA:30% demineralized FDBA) that is hydrated for 5 minutes in either sterile saline (control group) or a 4mg/ml dexamethasone solution (test group).

SECONDARY OUTCOMES:
Ridge Width | Baseline to 16 weeks (±2 weeks)
  Measurement of change in ridge width after healing
Buccal Ridge Height | Baseline to 16 weeks (±2 weeks)
  Measurement of change in ridge height after healing
Lingual Ridge Height | Baseline to 16 weeks (±2 weeks)
  Measurement of change in lingual ridge height after healing

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Mealey, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health Science Center at San Antonio, School of Dentistry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be de-identified prior to being shared with other investigators that are not part of the study team. If the results of this study are published in a peer review journal, participants will not be identified.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion when the results are published in a peer review journal